CLINICAL TRIAL: NCT06814080
Title: Residual Gastric Content and GLP-1
Status: Recruiting | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 287139
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pre-op Gastric Emptying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 8 hour fasting: A standardized gastric scanning protocol will be used, and patients classified following a 3-point grading system based solely on qualitative sonographic assessment of the antrum in the supine and right lateral decubitus positions. A qualitative assessment of the residual gastric fluid volume will be performed, according to the three-point grading scale previously described by Perlas et al. Grade 0 was defined by the absence of visualization of any content into a flat antrum in both the supine and the right lateral decubitus positions. Grade 1 was defined by the appearance of fluid content in the right lateral decubitus position only, and Grade 2 was defined by the visualization of fluid content in both the supine and the right lateral decubitus positions.
- 10 hour fasting: A standardized gastric scanning protocol will be used, and patients classified following a 3-point grading system based solely on qualitative sonographic assessment of the antrum in the supine and right lateral decubitus positions. A qualitative assessment of the residual gastric fluid volume will be performed, according to the three-point grading scale previously described by Perlas et al. Grade 0 was defined by the absence of visualization of any content into a flat antrum in both the supine and the right lateral decubitus positions. Grade 1 was defined by the appearance of fluid content in the right lateral decubitus position only, and Grade 2 was defined by the visualization of fluid content in both the supine and the right lateral decubitus positions.
- 12 hour fasting: A standardized gastric scanning protocol will be used, and patients classified following a 3-point grading system based solely on qualitative sonographic assessment of the antrum in the supine and right lateral decubitus positions. A qualitative assessment of the residual gastric fluid volume will be performed, according to the three-point grading scale previously described by Perlas et al. Grade 0 was defined by the absence of visualization of any content into a flat antrum in both the supine and the right lateral decubitus positions. Grade 1 was defined by the appearance of fluid content in the right lateral decubitus position only, and Grade 2 was defined by the visualization of fluid content in both the supine and the right lateral decubitus positions.

SUMMARY:
Studies have shown that even following the fasting guideline, patients on GLP-1 still have residual gastric content which increases their risk of aspiration during anesthesia. We aim to investigate the prevalence of full stomachs following different fasting times.

DETAILED DESCRIPTION:
Glucagon-like peptide-1 (GLP-1) receptor agonists have become increasingly popular as both diabetic and weight loss therapies. One effect of this class of medication is delayed gastric emptying, which may impact the risk of aspiration during anesthesia delivery. Some of them have a very long half-life of approximately one week. Thus, it takes approximately five weeks to achieve its steady-state concentration, and just as long for its effects to terminate after stopping the drug.

As a standard of care, patients are allowed to drink up to 2 hours and to eat up to 8 hours before surgery. Studies have shown that even following the fasting guideline, patients still have residual gastric content which increases their risk of aspiration during anesthesia. Since stopping these drugs for a long time is not practical as it is going to disrupt their glycemic control and reverse the weight loss, we propose to test extending the fasting time.

We aim to investigate the prevalence of full stomachs following different fasting times.

patients will be assigned to one of three groups: Group 1(G1) with 8-hour fasting, Group 2 (G2) with 10-hour fasting, and Group 3 (G3) groups with 12-hour fasting

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 yr. ASA physical status I- III Elective surgery

Exclusion Criteria:

* Pregnancy
* History of upper gastrointestinal disease or previous surgery on the esophagus, stomach or upper abdomen;
* Documented abnormalities of the upper gastrointestinal tract such as gastric tumors; recent upper gastrointestinal bleeding (within the preceding 1 month).
* Medicines that may delay gastric emptying (e.g., anticholinergic agents, opioid)
* ASA class IV or above
* Unable to understand English
* Cardiac cases with low ejection fraction
* Elderly patients above 65 years of age
* Liver or renal transplant cases
* Type 1 diabetes Patients on insulin or sulphonylurea medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects on GLP-1 scheduled for elective surgery will be screened for recruitment. We will find prospective subjects via medical records review or through our preoperative evaluation team which is a standard of care and then contact the patients about the study. Subjects enrolled in the study will be treated as per normal practice for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of full stomach or residual gastric content in the 3 groups | 8 hours
  Empty stomach when no content or clear liquids are visibly inferior to 1.5ml/kg. Full stomach includes the visualization of solids on gastric ultrasonography or a volume of clear liquids greater than 1.5ml/kg.
Prevalence of full stomach or residual gastric content in the 3 groups | 10 hours
  Empty stomach when no content or clear liquids are visibly inferior to 1.5ml/kg. Full stomach includes the visualization of solids on gastric ultrasonography or a volume of clear liquids greater than 1.5ml/kg.
Prevalence of full stomach or residual gastric content in the 3 groups | 12 hours
  Empty stomach when no content or clear liquids are visibly inferior to 1.5ml/kg. Full stomach includes the visualization of solids on gastric ultrasonography or a volume of clear liquids greater than 1.5ml/kg.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No